CLINICAL TRIAL: NCT05523401
Title: Acute Effects of 2C-B Compared With MDMA and Psilocybin in Healthy Subjects
Acronym: 2C-B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BASEC 2022-00355
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — 2-(4-bromo-2,5-dimethoxyphenyl)ethylamine; N-Methyl-3,4-methylenedioxyamphetamine; Psilocybin

STUDY DESIGN:
Intervention Model Description: 6-period random order, placebo-controlled, double-blind, cross-over study with five active substance conditions and placebo:
  1. 2C-B (10 mg), 2. 2C-B (20 mg), 3. 2C-B (30 mg), 4. MDMA (125 mg), 5. Psilocybin (25 mg), 6. Placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 10 mg 2C-B (Experimental): 2C-B (10 mg)
  Interventions: Drug: 4-bromo-2,5-dimethoxyphenethylamine (10 mg)
- 20 mg 2C-B (Experimental): 2C-B (20 mg)
  Interventions: Drug: 4-bromo-2,5-dimethoxyphenethylamine (20 mg)
- 30 mg 2C-B (Experimental): 2C-B (30 mg)
  Interventions: Drug: 4-bromo-2,5-dimethoxyphenethylamine (30 mg)
- 125 mg MDMA (Active Comparator): MDMA (125 mg)
  Interventions: Drug: 3,4-methylenedioxymethamphetamine
- 25 mg Psilocybin (Active Comparator): Psilocybin (25 mg)
  Interventions: Drug: Psilocybin
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 4-bromo-2,5-dimethoxyphenethylamine (10 mg) — A low dose of 10 mg 2C-B will be administered.
  Other Names: 2C-B
  Arms: 10 mg 2C-B
Drug: 4-bromo-2,5-dimethoxyphenethylamine (20 mg) — A medium dose of 20 mg 2C-B will be administered.
  Other Names: 2C-B
  Arms: 20 mg 2C-B
Drug: 4-bromo-2,5-dimethoxyphenethylamine (30 mg) — A high dose of 30 mg 2C-B will be administered.
  Other Names: 2C-B
  Arms: 30 mg 2C-B
Drug: 3,4-methylenedioxymethamphetamine — A moderate dose of 125 mg MDMA will be administered.
  Other Names: MDMA
  Arms: 125 mg MDMA
Drug: Psilocybin — A moderate dose of 25 mg psilocybin will be administered.
  Arms: 25 mg Psilocybin
Other: Placebo — Placebo (Mannitol)
  Arms: Placebo

SUMMARY:
4-bromo-2,5-dimethoxyphenethylamine (2C-B) is a psychoactive substance with reportedly similar acute effects to both the prototypical empathogen 3,4-methylenedioxymethamphetamine (MDMA, Ecstasy) and the classic psychedelic substance psilocybin (contained in "magic, hallucinogenic mushrooms"). Pharmacologically, MDMA mainly releases serotonin (5-HT) via the serotonin transporter (SERT) and psilocybin mainly acts as direct agonist at 5-HT2A receptors. 2C-B interacts with both the 5-HT2A receptor and SERT which is in line with its reported mixed effects profile. However, scientific studies are lacking. There is an increased interest in psychiatric research on the therapeutic properties of MDMA and psilocybin and also on mixed empathogenic-psychedelic substances.

DETAILED DESCRIPTION:
2C-B is a phenethylamine and belongs to the so-called 2C drugs, a group of novel psychoactive substances (NPS) with some structural similarity to the classic psychedelic mescaline. 2C-B is relatively widely used as recreational substance often replacing or mimicking classic substances such as LSD or MDMA. 2C-B also ranks high among the substances found as substitutes or adulterants of tablets sold as MDMA or Ecstasy. Users report that 2C-B has similar acute effects to MDMA when used at low (5-10 mg) and medium doses (10-25 mg) and more psychedelic effects when used at a high doses (25-40 mg). Additionally, in two open labeled studies the effects have been defined by the researchers as entactogenic (MDMA-like) with psychedelic/hallucinogenic properties when administering 20 mg and on the other hand as psychedelic-psychostimulant like when administering a mean dose of 16 mg (4 used 10 mg, 5 used 15 mg and 7 used 20 mg). Subjective effects peaked at 1-2h and lasted 5h.

The 2C drugs act mainly as agonists on the 5-HT2A receptor very similar to classic psychedelics like LSD or psilocybin. Furthermore, 2C-B may interact with monoaminergic systems more similar to MDMA and may share some empathogenic or even stimulant-type actions. 2C-B also inhibits the SERT similar to MDMA, however, only at low potency in vitro. Thus, taken together, the pharmacology of 2C-B in vitro is somewhat inconclusive but would be consistent with both MDMA- and psychedelic-type actions in vivo in humans. Increases in blood pressure and heart rate are moderate and regarded as lower than those of MDMA. No severe cases were observed. The safety profile of 2C-B is considered to be similar to MDMA.

Psilocybin is a classic serotonergic psychedelic. Psilocybin is a prodrug which is activated to psilocin within the body. The psychoactive action of psilocin primarily involves an interaction with the serotonin 5-HT2A receptor. Currently, psilocybin is the most investigated psychedelic substance among the classic psychedelics. In particular, there are high hopes of using psilocybin in patients with treatment resistant major depression and pharmaceutical companies are currently conducting phase III studies.

MDMA is an amphetamine derivative which, unlike prototypical amphetamines, predominantly enhances serotonergic neurotransmission via release of 5-HT through the SERT and it less potently also releases dopamine and norepinephrine through the dopamine transporter (DAT) and norepinephrine transporter (NET), respectively. Furthermore, MDMA is known to trigger oxytocin release which may contribute to its effects to increase trust, prosociality, and enhanced empathy and is therefore referred to as an "entactogen" or "empathogen". Being granted as a "breakthrough therapy" by the FDA, MDMA is currently investigated in substance-assisted psychotherapy for treatment of PTSD.

By using a placebo-controlled double-blind cross-over design the study will provide insight into the effects profiles of recreationally used psychoactive substances relevant for psychiatric research. Therefore the study will compare the acute subjective, physiological and endocrine effects of low (10 mg), medium (20 mg) and high (30 mg) doses of 2C-B with standard doses of MDMA (125 mg) and psilocybin (25 mg) in healthy subjects.

Finally, the study will also allow to newly directly compare MDMA and psilocybin effects at representative doses and within the same subjects which will provide for a better characterization of these substances increasingly used in psychiatric research.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 and 65 years.
* Sufficient understanding of the German language.
* Understanding the procedures and the risks that are associated with the study.
* Participants must be willing to adhere to the protocol and sign the consent form.
* Participants must be willing to refrain from taking illicit psychoactive substances during the study.
* Participants must be willing to drink only alcohol-free liquids and no coffee, black or green tea, or energy drink after midnight of the evening before the study session, as well as during the study day.
* Participants must be willing not to drive a traffic vehicle or to operate machines within 48 h after substance administration.
* Women of childbearing potential must have a negative pregnancy test at the beginning of the study. Pregnancy tests are repeated before each study session.
* Women of childbearing potential must be willing to use double-barrier birth control.
* Body mass index between 18-29kg/m2

Exclusion Criteria:

* Chronic or acute medical condition, including a history of seizures.
* Current or previous major psychiatric disorder (e.g. psychotic disorders, mania / hypomania, anxiety disorders).
* Psychotic or bipolar disorder in first-degree relatives, not including psychotic disorders secondary to an apparent medical reason, e.g. brain injury, dementia, or lesions of the brain.
* Hypertension (SBP>140/90 mmHg) or hypotension (SBP<85 mmHg)
* Ilicit substance use (with the exception of cannabis) more than 20 times or any time within the previous two months
* Pregnant or nursing women.
* Participation in another clinical trial (currently or within the last 30 days).
* Use of medications that may interfere with the effects of the study medications (any psychiatric medications and any medication with known to interact with the study substances).
* Tobacco smoking (>10 cigarettes/day).
* Consumption of alcoholic drinks (>20 drinks / week).
* Body weigt < 45 kg.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Acute subjective effects I | 18 months
  5 Dimensions of Altered States of Consciousness (5D-ASC) consisting of 94 items to be rated on a visual analog scale (0-100 mm), with higher values indicating stronger effects with higher scores representing more intense effects.
  Assessed once at the end of the session, 9h after substance administration.

SECONDARY OUTCOMES:
Acute subjective effects II | 18 months
  Visual Analog Scale (VAS) will be repeatedly used to assess subjective alterations in consciousness over time. Scales will be administered 14 times throughout the study day.
Acute subjective effects III | 18 months
  The Adjective Mood Rating Scale (AMRS) assesses the occurrence and intensity of 60 moods on a 4-point Likert scale ranging from "not at all" to "extremely". It will administred 4 times throughout the study day.
Autonomic effects I | 18 months
  Assessed 15 times on each study day via systolic and diastolic blood pressure.
Autonomic effects II | 18 months
  Assessed 15 times on each study day via heart rate.
Autonomic effects III | 18 months
  Assessed 15 times on each study day via tympanic body temperature.
Plasma levels of 2C-B, MDMA, and psilocybin | 18 months
  Assessed 14 times on each study day via blood samples.
Plasma levels of oxytocin | 18 months
  Assessed 4 times on each study day via blood samples.
Plasma levels of Brain-derived neurotropic factor (BDNF) | 18 months
  Assessed 4 times on each study day via blood samples.
Adverse effects | 18 months
  The list of complaints (LC) consists of 66 items, yielding a global score measuring physical and general discomfort. The LC list is administered before (describing the last 24 h as baseline) and after substance administration at the end of the study day describing the acute adverse effects.
Urine Recovery | 18 months
  Urine samples will be collected after 2C-B / psilocybin / MDMA / placebo administration (0- 9h).
States of Consciousness Questionnaire | 18 months
  Assesses the emergence and intensity of phenomenons occurring in altered states of consciousness on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely"). The scale will be administered once, 9 h after drug administration.
Spiritual Realms Questionnaire | 18 months
  Assesses the spiritual phenomenons elicited by psychedelic substances through 11 main questions to be answered on a total of 65 sub-ordered 100mm visual analog scales. The scale will be administered once, 9 hours after substance administration.
Psychological Insight Questionnaire | 18 months
  Assesses the degree of psychological insight caused by a psychedelic experience through 14-items to be answered on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely"). The PIQ will be administered once on each study day, 9 hours after substance administration.
NEO-Five-Factor-Inventory (NEO-FFI) | Baseline
  The NEO-FFI is a self-description questionnaire with 60 items for the measurement of the "big five": neuroticism, extraversion, openness, agreeableness, and consciousness. It uses a 5-point Likert scale ranging from "completely disagree" to "fully agree".
Freiburger Personality Inventory (FPI-R) | Baseline
  The FPI-R version comprises 138 items and covers 12 dimensions of personality: life satisfaction, social orientation, performance orientation, inhibition, excitability, aggressiveness, stress, physical complaints, health concerns, openness, as well as the secondary factors according to Eysenck's Extraversion and Emotionality (Neuroticism). It uses a 2-point scale ("true" and "not true").
Saarbrücker Personality Questionnaire (SPF) | Baseline
  The SPF defines empathy as the "reactions of one individual to the observed experiences of another." It assesses 28- items on a 5-point Likert scale ranging from "Does not describe me well" to "Describes me very well". The measure has 4 subscales (Perspective Taking, Fantasy, Empathic Concern, Personal Distress) each made up of 7 different items.
HEXACO personality inventory | Baseline
  The HEXACO personality inventory is a six-dimensional model of human personality with 100 items.The six factors are: Honesty-Humility, Emotionality, Extraversion, Agreeableness, Conscientiousness and Openness to Experience.
Defense Style Questionnaire (DSQ-40) | Baseline
  The DSQ-40 can provide scores for 20 individual defenses, and scores for the three factors "mature", "neurotic", and "immature". Each item is evaluated on a scale from 1 to 9, where "1" indicates "completely disagree" and "9" indicates "fully agree".

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland